CLINICAL TRIAL: NCT00535717
Title: Role of Uttarbasti in the Management of Mutra Marga Sankoch (Urethral Stricture)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maharashtra University of Health Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUHS RIA
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Urethral Stricture
Keywords: Urethral stricture; Ayurvedic treatment; mutra marg sankoch; uttarbasti; Sesame oil; Honey; Rock salt
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: uttarbasti (per urethral administration of medicated oil )

SUMMARY:
Uttarbasti is per urethral administration of medicated oil which has been recommended by Sushrut for urinary track disorders.

As far as conventional surgery is concerned urethral stricture still remains a challenge due to post procedural high recurrences and complications

Uttarbasti being almost non invasive, with minimum recurrences and most economical, easy to practice OPD procedure, can be the treatment of choice in the management of urethral stricture.

ELIGIBILITY:
Inclusion Criteria:

* K/C/O Urethral Stricture of either sex and from all age groups.

Exclusion Criteria:

* With acute UTI.
* DM.
* Neoplasms of lower urinary tract
* BEP.
* With impacted calculus in urethra and bladder neck.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra H Amilkanthwar, M.D.(Ayu.), Principal Investigator — Maharashtra university of health sciences, Nashik (INDIA)